CLINICAL TRIAL: NCT00645333
Title: Phase I/II Trial of MK-0752 Followed by Docetaxel in Locally Advanced or Metastatic Breast Cancer: A Study by the Stem Cell Clinical Consortium
Brief Title: Phase I/II Study of MK-0752 Followed by Docetaxel in Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Baylor College of Medicine (Other); Ohio State University (Other); Dana-Farber Cancer Institute (Other); Weill Medical College of Cornell University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ann Schott, MD, Principal Investigator, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.119
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; Phase I clinical trial; cancer stem cells; agents with other mechanisms of action; Notch inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — 3-(4-((4-chlorophenyl)sulfonyl)-4-(2,5-difluorophenyl)cyclohexyl)propanoic acid; Docetaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-0752, Docetaxel, Pegfilgrastim (Experimental): MK-0752, Docetaxel, Pegfilgrastim in combination with escalating doses of MK-0752
  Interventions: Drug: MK-0752, Docetaxel, Pegfilgrastim

INTERVENTIONS:
Drug: MK-0752, Docetaxel, Pegfilgrastim — MK-0752 in escalating doses of 300, 450, 600, and 800 mg given orally on days 1-3, followed by docetaxel 80 mg/m2 day 8 and pegfilgrastim 6 mg SQ on day 9
  Other Names: Taxotere; Neulasta

SUMMARY:
New and better therapies for locally advanced and metastatic breast cancer are needed because, even if standard treatment is successful in shrinking the cancer, there is still a high chance that the cancer will recur. Recent research suggests that breast tumors have a small number of cells in them that are "breast cancer stem cells", which are very resistant to standard treatment. It is thought that the reason that many patients cannot be cured of their breast cancers is that the stem cells are unable to be killed and remain in the body after standard treatment. Laboratory research has shown that a new drug, MK-0752, can target stem cells and prevent tumor recurrences when the drug is combined with docetaxel, a chemotherapy drug commonly used to treat breast cancer.

We know that MK-0752 is safe when given by itself to people. We do not know if treatment with MK-0752 and docetaxel combined is safe or if it will kill "breast cancer stem cells" in people with breast cancer. This clinical trial is being done to determine the safety of several doses of MK-0752 in combination with docetaxel. Preliminary data about the effectiveness of MK-0752 in combination with docetaxel will be collected. Also, tumor biopsy samples will be taken from some patients who have tumors that can be easily biopsied. The samples will be used to perform research tests to help determine if the "breast cancer stem cells" are being killed by the drug combination.

DETAILED DESCRIPTION:
Purpose-Accumulating evidence supports the existence of breast cancer stem cells (BCSCs), which are characterized by their capacity to self-renew and divide indefinitely, and resistance to conventional therapies. The Notch pathway is important for stem cell renewal, and is a potential target for BCSC-directed therapy. Experimental Design-Using human breast tumorgraft studies, we evaluated the impact of gamma secretase inhibitors (GSI) on the BCSC population and the efficacy of combining GSI with docetaxel treatment. The mouse experimental therapy paralleled a concurrent clinical trial in advanced breast cancer patients, designed to determine the maximally tolerated dose of the GSI, MK-0752, administered sequentially with docetaxel, and to evaluate BCSC markers in serial tumor biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with metastatic (Stage IV) breast cancer, or with locally advanced breast cancer (Stages IIIA > 10 cm, or Stages IIIB and IIIC) that did not respond to first-line anthracycline-based chemotherapy, for whom docetaxel is a recommended therapy
* Presence of measurable or evaluable disease
* Adequate organ function
* Ability to swallow intact study drug capsules
* Zubrod Performance Status of 0-1 with at least a 3 month life expectancy
* Appropriate time must have elapsed since prior anti-neoplastic therapy with resolution of acute toxicity

Exclusion Criteria:

* Concurrent treatment with hormonal therapy intended to treat cancer
* Radiotherapy within 7 days prior to first dose
* Symptomatic central nervous system, and/or epidural metastases or symptomatic carcinomatous meningitis or with radiation treatment completed within the past 8 weeks
* Serious comorbid illness which will limit the ability of the patient to safely receive anticancer treatment
* Patients who are pregnant or nursing
* Confounding factors present to provide misinterpretation of data (i.e., concurrent malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Schott, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Schott AF, Landis MD, Dontu G, Griffith KA, Layman RM, Krop I, Paskett LA, Wong H, Dobrolecki LE, Lewis MT, Froehlich AM, Paranilam J, Hayes DF, Wicha MS, Chang JC. Preclinical and clinical studies of gamma secretase inhibitors with docetaxel on human breast tumors. Clin Cancer Res. 2013 Mar 15;19(6):1512-24. doi: 10.1158/1078-0432.CCR-11-3326. Epub 2013 Jan 22. PMID 23340294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects included men or women with metastatic (Stage IV)breast cancer, or with locally advanced breast cancer (Stages IIIA> 10cm, or stages IIIB and IIIC) that did not respond to first-line anthracycline-based chemotherapy.
Pre-assignment Details: There must b at least a 6 month interval since prior taxane therapy.
Groups:
- MK-0752 and Docetaxel: MK-0752 in escalating doses, orally days 1-3, followed by docetaxel 80 mg/m2 IV on day 8, and pegfilgrastim 6mg SQ day 9. Cycle repeated every 21 days.
Period: Overall Study
Arm/Group | MK-0752 and Docetaxel
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MK-0752 and Docetaxel
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Metastatic sites (multiple sites possible) [Number; unit: Participants] — Metastatic sites at baseline. Patients may have more than one metastatic site at baseline and therefore the total numbers for all categories (all metastatic sites) may be greater than the overall number of baseline participants.
  Participants
    Bone | 12
    Lung/Pleura | 16
    Liver | 13
    Lymph Nodes | 11
    Skin | 5
    Other | 7
Number of Metastatic Sites [Number; unit: participants]
  0 | 4
  1 | 6
  2 | 6
  >=3 | 14
Tumor Hormone Receptor Status [Number; unit: Participants]
  ER positive/or PgR positive | 18
  ER negative and PgR negative | 12
HER-2/neu status [Number; unit: Participants]
  Negative | 28
  Positive | 2
Prior Therapy For Metastatic Disease [Number; unit: Participants] — Prior therapy for metastatic disease. Patients may have had more than one prior therapy and therefore the total numbers for all categories (all prior therapies) may be greater than the overall number of baseline participants.
  Participants
    None | 7
    Chemotherapy | 7
    Hormonal Therapy | 0
    Chemotherapy and Hormonal Therapy | 16
Number of Prior Metastatic Chemotherapy Regimens [Number; unit: Participants] — Number of prior metastatic chemotherapy regimens. Patients may have more than one prior metastatic chemotherapy regimen and therefore the total numbers for all categories (all prior metastatic chemotherapy regimens) may be greater than the overall number of baseline participants.
  Participants
    0 | 7
    1 | 2
    2+ | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: The number of DLTs experienced by participants within the first 21 days.
  DLTs were defined as toxicities possibly, probably, or definitely related to the study drug observed during the first 2 cycles (first 42 days) as follows:
  1. Non-hematologic toxicity Grade ≥3 by the NCI CTCAE version 3.0.
  2. ANC<1000 for more than 7 days despite use of pegfilgrastim.
  3. Platelet count <25,000 for more than 7 days, or associated with bleeding, or less than 10,000 at any time.
Time Frame: first 21 days
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | MK-0752 and Docetaxel
Number analyzed (Participants) | 30
Dose Limiting Toxicities | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The Maximum Tolerated Dose (MTD) for MK-0752 will be determined. Dose levels were: Level 1: 300 mg MK-0752 by mouth days 1-3; Level 2: 450 mg MK-0752 by mouth days 1-3; Level 3: 600 mg MK-0752 by mouth days 1-3; Level 4: 800 mg MK-0752 by mouth days 1-3.
Time Frame: Up to 3 years
Measure: Number; unit: mg
Arm/Group | MK-0752 and Docetaxel
Number analyzed (Participants) | 30
mg | 600

ADVERSE EVENTS:
Time Frame: During therapy and for 30 days after therapy completion
Groups:
- MK-0752: MK-0752 in escalating doses, orally days 1-3, followed by docetaxel 80 mg/m2 IV on day 8, and pegfilgrastim 6mg SQ day 9. Cycle repeated every 21 days.
Arm/Group | MK-0752
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0752 (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 1 (1)
Device related infection (Infections and infestations) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand-and-foot syndrome (Nervous system disorders) | 1 (1)
Hypersensitivity (General disorders) | 2 (6)
Immune system disorder (Immune system disorders) | 1 (1)
Infection, Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0752 (N=30)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alanine aminotransferase increased (Investigations) | 5 (9)
Alkaline phosphatase increased (Investigations) | 8 (12)
Allergic reaction (Immune system disorders) | 4 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 7 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cardiac Arrhythmia - Other (Specify) (Cardiac disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Depression (Psychiatric disorders) | 2 (2)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 10 (12)
Dry eye syndrome (Eye disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 20 (26)
Fever (General disorders) | 7 (10)
GI - Other (Specify) (Gastrointestinal disorders) | 2 (2)
Hand-and-foot syndrome (Nervous system disorders) | 7 (10)
Headache (Nervous system disorders) | 4 (5)
Hemoglobin (Blood and lymphatic system disorders) | 11 (16)
Hot flashes (Vascular disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (19)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (10)
Hypokalemia (Metabolism and nutrition disorders) | 9 (12)
Insomnia (Psychiatric disorders) | 5 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Leukocytes (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 4 (5)
Nail changes (Skin and subcutaneous tissue disorders) | 10 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (17)
Pain - Other (General disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (13)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (7)
Skin infection (Infections and infestations) | 3 (3)
Sweating (General disorders) | 2 (2)
Taste alteration (Nervous system disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Urinary tract infection (Renal and urinary disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6)
Watering eyes (Eye disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No